CLINICAL TRIAL: NCT01293578
Title: Translating Information on Comparative Effectiveness Into Practice (TRICEP)
Brief Title: Study to Test Use of a Decision Aid in a Clinical Visit to Help Patients Choose a Diabetes Medication
Acronym: TRICEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10-006952
Record Dates: First submitted 2011-02-01; First posted 2011-02-10 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Decision Aids; Shared Medical Decision Making; Patient Education; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Clinicians will present diabetes medication options to patients, in their usual way.
- Diabetes Medication Decision Aid (Experimental): In the decision aid arm, clinicians will use the diabetes medication decision aid cards (if they choose) when discussing diabetes medication options with their patients.
  Interventions: Other: Diabetes Medication Choice Cards

INTERVENTIONS:
Other: Diabetes Medication Choice Cards — Clinician uses the Diabetes Medication Choice Cards to inform and engage patient in discussing the issues they find relevant in choosing a new diabetes medication.
  Arms: Diabetes Medication Decision Aid

SUMMARY:
The goal of this study is to test the relative merits of a decision aid for diabetes medications that we have developed - Diabetes Medication Choice Cards- versus usual care in translating comparative effectiveness research (CER) into real world clinics. This study will involve about 20 primary care practice sites affiliated with Mayo Health System, Park Nicollet, or Hennepin County Medical Center. There will be no recruiting done at the Mayo Clinic.

DETAILED DESCRIPTION:
To conduct a cluster-randomized practical trial to evaluate the impact of our decision aid (Diabetes Medication Choice Cards) versus usual care as strategies to translate CER into practice among patients with poorly controlled diabetes in need of drug intensification (Hemoglobin Alc (HbA1c) > 7.3%). Patient outcomes including reaching glycemic control target (HbA1c less than or equal to 7.3%), medication choice and adherence, satisfaction and knowledge. From the physician perspective, we will be measuring physician adoption and satisfaction with the decision aid.

To identify, describe, and explain factors that promote or inhibit the uptake of complex interventions such as decision aids in practices participating in the trial.

To conduct an exploratory analysis of the ability of patients to adhere to the medications chosen while exploring the factors that enable or hinder the patients' ability to incorporate these medications into their routine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Have a diagnosis of Type 2 diabetes mellitus and on diabetes medication
* Have a diagnosis of Type 2 diabetes mellitus for 1 year or more if not currently on diabetes medication
* Recognize their primary care provider as their main diabetes care provider
* Use 0, 1, 2, or 3 oral hypoglycemic agents
* Have a recent HbA1c measure (within 12 months) of greater than 7.3, with priority to patients with rising HbA1c levels.

Exclusion Criteria:

* Not available for follow-up for 12 months after study visit.
* Unable to read and speak English.
* Has major barriers to providing written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction and knowledge | baseline to 12 months
  Primary outcome is to evaluate the impact of our decision aid (Diabetes Medication Choice Cards) versus usual care as strategies to translate CER into practice among patients with poorly controlled diabetes in need of drug intensification (Hemoglobin A1c (HbA1c) > 7.3%). Patient outcomes include satisfaction with use of the decision aid and knowledge, compared to the control, usual care group (by written survey at point of care and follow-up).

SECONDARY OUTCOMES:
Physician adoption and satisfaction with the decision aid. | baseline to 12 months
  Brief post-visit surveys will be completed by the clinicians, directly following clinical visit.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Albert Lea Medical Center, Albert Lea, Minnesota
  - Mayo Clinic Kasson, Kasson, Minnesota
  - Mayo Clinic Health System- Immanual St. Joseph's, Mankato, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- [Result] Kunneman M, Branda ME, Ridgeway JL, Tiedje K, May CR, Linzer M, Inselman J, Buffington ALH, Coffey J, Boehm D, Deming J, Dick S, van Houten H, LeBlanc A, Liesinger J, Lima J, Nordeen J, Pencille L, Poplau S, Reed S, Vannelli A, Yost KJ, Ziegenfuss JY, Smith SA, Montori VM, Shah ND. Making sense of diabetes medication decisions: a mixed methods cluster randomized trial using a conversation aid intervention. Endocrine. 2022 Feb;75(2):377-391. doi: 10.1007/s12020-021-02861-4. Epub 2021 Sep 9. PMID 34499328
- [Derived] Montori VM, Ruissen MM, Branda ME, Hargraves IG, Kunneman M. Problem-based shared decision making: The role of canonical SDM steps. Health Expect. 2023 Feb;26(1):282-289. doi: 10.1111/hex.13654. Epub 2022 Nov 29. PMID 36448245
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials